CLINICAL TRIAL: NCT02603978
Title: Examining the Efficacy of Interventions for Sexual Assault: A Preliminary Randomized Controlled Trial
Brief Title: Interventions for Sanctioned Ohio University Students
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ohio University (Other)
Collaborators: American Psychological Foundation (Other)
Responsible Party: Principal Investigator, Ryan Shorey, Assistant Professor of Psychology, Ohio University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 15F018
Record Dates: First submitted 2015-11-06; First posted 2015-11-13 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Wait-list (No Intervention): This arm will receive no intervention for the first 6 months. At the conclusion of the 6-month period, this group will receive a brief alcohol intervention
- Brief Alcohol Intervention (Active Comparator): This arm will receive a brief (2-hour) alcohol intervention based on motivational interviewing
  Interventions: Behavioral: BASICS
- Bystander and Social Norms Intervention (Active Comparator): This arm will receive a brief (2-hour) bystander and social norms intervention designed to increase healthy sexual behaviors
  Interventions: Behavioral: Bystander and Social Norms
- Combined Alcohol and Bystander Intervention (Active Comparator): This arm will receive a combined (4-hour) alcohol and bystander/social norms intervention to target both alcohol and sexual behavior
  Interventions: Behavioral: Combined BASICS and Bystander

INTERVENTIONS:
Behavioral: BASICS — A 2-hour group intervention focused on reducing alcohol use with the use of motivational interviewing
  Arms: Brief Alcohol Intervention
Behavioral: Bystander and Social Norms — A 2-hour group intervention focused on increasing healthy sexual behaviors and prosocial bystander behavior
  Arms: Bystander and Social Norms Intervention
Behavioral: Combined BASICS and Bystander — A 2-session, 4-hour group that consists of both BASICS and the Bystander intervention
  Arms: Combined Alcohol and Bystander Intervention

SUMMARY:
The purpose of this study is to determine whether (a) a brief alcohol intervention, (b) a brief bystander and social norms intervention, or (c) a brief alcohol and a brief bystander and social norms intervention are effective at reducing alcohol use and sexual-related behaviors among college men mandated to receive an alcohol intervention by their university.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 or older; must be an ohio university student; must be male; must be sanctioned to receive an alcohol intervention by Ohio University

Exclusion Criteria:

* Under the age of 18; not attending the main Ohio University campus (Athens)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
The Alcohol Use Disorders Identification Test | 6 months post-intervention
  A self-report measure that examines alcohol use and problems. This measure produces one total score that is interpreted as "alcohol use and problems."
Bystander Behavior Scale | 6 months post-intervention
  A self-report measure that examines opportunities and engagement in prosocial bystander behavior. A single total score is obtained by calculating the percentage of times individuals engaged in bystander behavior based on the number of opportunities they had for such behavior.